CLINICAL TRIAL: NCT00255957
Title: Clinical Trial to Study the Effects of HES on Coagulation, Hemorehology and Kinetics Comparing Two Different Products.
Brief Title: Influence of Hydroxyehtyl Starch (HES) on Hemorehology, Coagulation and Elimination Kinetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nizam's Institute of Medical Sciences University, India (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIMS HES 1
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2006-04-19 (Estimated); Status verified 2005-11

CONDITIONS: Stroke Patients Presenting Within 24 Hrs of Onset of Symptoms
Keywords: Stroke, HES, Coagulation, Kinetics, Hemorehology
MeSH Terms: conditions — Stroke; Hypereosinophilic Syndrome; Thrombosis

INTERVENTIONS:
Drug: HES administration
Drug: Hydroxy Ethyl Starch administration to stroke patients

SUMMARY:
The use of HES has been found clinically to improve patients with stroke if administered within a window period by means of hemodilution to improve rehology. We propose to see the effects of long term administraion of HES in the amounts required for treating stroke patients and study the effects on the kinetics of HES, its effects on coagulation and hemorheology.

DETAILED DESCRIPTION:
Patients with stroke benefit with hemodilution when administered HES in a window period and continued for a period of 10 days. Hemodilution improves the hemorheology and thus possibly preserves the cerebral tissues in the penumbra regions of affected vessels.

We propose to see the effects of prolonged administration of HES from different makes and study the kinetics, hemorehology and coagulation parameters by TEG as there is no literature on kinetics and coagulation follwing prolonged use in stroke patients and also study their neurological outcomes.

Patients presenting to the Emergency department or outpatient department within 24 hrs of manifestation of symptoms will be recruited to the study after taking informed consent in a language the patients/ family understand by the study personnel identified and authorized to do the same.

The patients will then be randomly allocated to receive HES of either make for 10 day with 10 patients in each group.

The randomization is by random number generation by computer.

The product is blinded to the patient and observer by black cover with only the label A OR B of each group.

Blood Samples will be drawn at time of randomization, after 3, 5 and 10 days for rehological, coagulation effects and kinetics of HES, stored as per requirements and analyzed. Routine biochemical tests as prescribed by the physician will be undertaken as required.

Satistical analysis of data will be done by SPSS.

ELIGIBILITY:
Inclusion Criteria:

Age 18 - 70 yrs Clinical diagnosis of ischemic stroke No marked spontaneous improvement of symptoms before randomization Written informed consent from nearest relative.

-

Exclusion Criteria:

Pregnancy Allergy to HES Severe impairment of consciousness Previous stroke with persistent ipsilateral deficits. Seizure at stroke onset. Intracranial neoplasm or AV malformation. Cardiac insufficiency or pulmonary edema Myocardial infarction during the previous 3 months or unstable angina. Severe dehydration Coagulation disorders. Uncontrolled Hypertension. Laboratory findings reflecting severe anemia, renal insufficiency, thrombocytopenia or hepatic insufficiency.

Participation in another clinical trial within the previous 2 months or concurrent treatment with any other experimental drug.

SECONDARY EXCLUSION CRITERIA.

Cerebral CT at enrolment showing intracranial hemorrhage of any degree-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-10; Study Completion 2006-03

PRIMARY OUTCOMES:
Patients discharged from hospital

SECONDARY OUTCOMES:
Coagulation, rehology and kinetics measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Ramachandran Gopinath, MD,DA,FFARCSI, Principal Investigator — NIZAM'S INSTITUTE OF MEDICAL SCIENCES, PANJAGUTTA, HYDERABAD, INDIA